CLINICAL TRIAL: NCT02351817
Title: An Explorative Randomized Controlled Investigation Evaluating Newly Developed Ostomy Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP256
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Ileostomy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline - Test A - Test B (Experimental): Three period investigation. First each subject tests baseline product, then Test A and finally Test B.
  Baseline product: the subject's usual product
  Test A: A newly developed 1-piece, open ostomy appliance for collecting feces
  Test B: A newly developed 1-piece, open ostomy appliance for collecting feces
  Interventions: Device: Test A; Device: Test B; Device: Baseline
- Baseline - Test B - Test A (Experimental): First each subject tests baseline product, then Test B and finally Test A.
  Baseline product: the subject's usual product
  Test A: A newly developed 1-piece, open ostomy appliance for collecting feces
  Test B: A newly developed 1-piece, open ostomy appliance for collecting feces
  Interventions: Device: Test A; Device: Test B; Device: Baseline

INTERVENTIONS:
Device: Test A — Ostomy appliance
Device: Test B — Ostomy appliance
Device: Baseline — Ostomy appliance

SUMMARY:
The primary objective of the investigation is to explore the acceptance of a newly developed adhesive.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent and letter of authority
* Be at least 18 years of age and have full legal capacity
* Be able to handle the products her/himself
* Have an ileostomy with a diameter between 10 and 30 mm
* Willing to follow the product change schedule (one change per day)
* Have had their ostomy for at least three months
* Willing to use 1 piece open ostomy products during the test period
* Must be able to use a custom cut product
* Have intact skin
* Negative result of a pregnancy test for women of childbearing age

Exclusion Criteria:

* Currently receiving or have within the past 2 months received radio- and/or chemotherapy
* Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/ injection) treatment
* Is pregnant or breastfeeding.
* Is participating in other interventional clinical investigations or have previously participated in this investigation
* Have a loop ileostomy
* Known hypersensitivity towards any of the test products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte Petersen Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline - Test A - Test B: First each subject tests baseline product, then Test A and finally Test B.
  Baseline product: the subject's usual product
  Test A: A newly developed 1-piece, open ostomy appliance for collecting feces
  Test B: A newly developed 1-piece, open ostomy appliance for collecting feces
Period: Baseline Period
Arm/Group | Baseline - Test A - Test B | Baseline - Test B - Test A
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Period 1
Arm/Group | Baseline - Test A - Test B | Baseline - Test B - Test A
Started | 5 | 5
Completed | 4 | 2
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Period: Period 2
Arm/Group | Baseline - Test A - Test B | Baseline - Test B - Test A
Started | 5 (Subjects who did not complete Period 1 as planned were allowed to continue to Period 2) | 5 (Subjects who did not complete Period 1 as planned were allowed to continue to Period 2)
Completed | 4 | 3
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Ileostomy opereated subjects
Groups:
- Overall Study Population: The investigation is a cross-over investigation therefore baseline data is presented for the overall population
Arm/Group | Overall Study Population
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Product Acceptance
Description: Product acceptance was measurement qualitatively by interviews exploring the factors and mechanisms affecting the acceptance. The interview questions were formulated in such a way that was not possible to quantify the number of subjects accepting the test products.
  There were problems with test product performance and handling and therefore the acceptance of the products was not high. Product preference was secondary endpoint, where the subjects were asked whether they preffered their own product over the test products. This endpoint is the best measure we have for mimiking product acceptance. However, we are aware subjects could accept a product without preferring it over own product and the preferrence result might therefore not be accurate.
  The result presented below shows how many subjects preferred Test A/Test B over own product
Time Frame: 7 days per test period
Population: One subject did not answer the preference question.
Measure: Number; unit: participants
Groups:
- Test A: How many subjects preferred Test A over own product
- Test B: How many subjects preferred Test B over own product
Arm/Group | Test A | Test B
Number analyzed (Participants) | 9 | 9
participants | 0 | 1

ADVERSE EVENTS:
Groups:
- Baseline: Adverse events reported by subjects testing Own product
- Test A: Adverse events reported by subjects testing Test A
- Test B: Adverse events reported by subjects testing Test B
Arm/Group | Baseline | Test A | Test B
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 3/10 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (N=10) | Test A (N=10) | Test B (N=10)
Common Cold with fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — not related to device
Peristomal skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pain from peristomal skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — not related to device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes